CLINICAL TRIAL: NCT04163107
Title: Combined Carfilzomib and Hydroxychloroquine in Patients With Relapsed/Refractory Multiple Myeloma - a Phase 1 Trial
Brief Title: Combined Carfilzomib and Hydroxychloroquine in Patients With Relapsed/Refractory Multiple Myeloma
Acronym: MYELOMA-HCQ
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019/922; 2019-000986-19 (EudraCT Number)
Record Dates: First submitted 2019-11-11; First posted 2019-11-14 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Multiple Myeloma
Keywords: Drug Therapy; Administration and Dosage; Hydroxychloroquine; Carfilzomib; Dexamethasone; Drug Therapy, Combination
MeSH Terms: conditions — Multiple Myeloma | interventions — Hydroxychloroquine; carfilzomib; Dexamethasone

STUDY DESIGN:
Intervention Model Description: A single arm, dose escalation study in two centers. 3+3 design in five dose levels.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination treatment of carfilzomib/dexamethasone/HCQ (Experimental)
  Interventions: Drug: Hydroxychloroquine; Drug: Carfilzomib Injection; Drug: Dexamethasone

INTERVENTIONS:
Drug: Hydroxychloroquine — All patients start with a 14 days run-in with monotherapy with hydroxychloroquine (HCQ) at their assigned dose level. Then they continue with 6 28-day cycles of HCQ/Carfilzomib/Dexamethasone. 3 patients at each dose level.
Drug: Carfilzomib Injection — All patients start with a 14 days run-in with monotherapy with hydroxychloroquine (HCQ) at their assigned dose level. Then they continue with 6 28-day cycles of HCQ/Carfilzomib/Dexamethasone. 3 patients at each dose level.
Drug: Dexamethasone — All patients start with a 14 days run-in with monotherapy with hydroxychloroquine (HCQ) at their assigned dose level. Then they continue with 6 28-day cycles of HCQ/Carfilzomib/Dexamethasone. 3 patients at each dose level.

SUMMARY:
Multiple myeloma (MM) is a neoplastic expansion of bone marrow plasma cells. Despite advances in treatment in recent years, MM is still a fatal disease. MM is characterized by the ability of malignant cells to produce large amounts of monoclonal immunoglobulin. The secretion of these immunoglobulins can be detected as the "M-protein" in serum, and the measurement of the M-component is used both for diagnosis and to evaluate treatment response and relapse. The high load of secreted proteins in MM cells requires a efficient way to clear these proteins from the cells and targeting protein degradation is an important therapeutic target in MM. This is today done by inhibiting the proteasome, one of the two central ways cells can degrade proteins, by drugs named proteasome inhibitors (including bortezomib, ixazomib and carfilzomib). Patients become resistant to these drugs, and it is therefore likely that myeloma cells also utilise another important system for protein degradation, called autophagy. Pre-clinical studies have shown that the combination of the proteasome inhibitor carfilzomib and the autophagy inhibitor hydroxychloroquine increases myeloma cell death and that hydroxychloroquine is able to reverse MM cell resistance to carfilzomib. This is the rationale for this study, where the investigators add the autophagy inhibitor hydroxychloroquine to a standard regime of carfilzomib and dexamethasone, to determine a maximum tolerated dose of this combination and to study tolerability.

ELIGIBILITY:
Inclusion Criteria:

Demographic and diagnosis

* A prior diagnosis of multiple myeloma according to International Myeloma Working Group (IMWG) criteria with documented disease progression in need of treatment at time of screening.

  - Must meet all of the following criteria:
* Patients must have received at least two prior therapies including bortezomib and an immunomodulatory agent (may include autologous bone marrow transplantation)
* Patients must not be refractory to carfilzomib
* Relapsed or progressive disease documented according to IMWG criteria
* Patients must have evaluable multiple myeloma with at least one of the following (assessed within 21 days prior to registration)
* Serum M-protein ≥ 10 g/L, or
* Urine M-protein ≥ 200 mg/24 hours
* Involved serum immunoglobulin free light chain (SFLC) > 100 mg/L AND abnormal kappa/lambda ratio
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Life expectancy ≥ 6 months

Laboratory:

* Absolute neutrophil count ≥ 1.0 x 109/L
* Hemoglobin ≥ 7 g/dL (with or without transfusion support)
* Platelets ≥ 50 x 109/L (with or without transfusion support)
* Total bilirubin ≤ 2 x upper limit of normal (ULN)
* Aspartate amino transferase/alanine amino transferase ratio (ASAT/ALAT) ≤ 2.5 x ULN
* Creatinine ≤ 2 x ULN

Concurrent conditions

* Left ventricular ejection fraction (LVEF) ≥ 40 % determined by 2D transthoracic echocardiogram (ECHO) or Multigated Acquisition Scan (MUGA)
* No baseline peripheral neuropathy ≥ grade 2
* No history of allergic reactions to compounds of similar chemical or biological composition to carfilzomib, dexamethasone or hydroxychloroquine, including Captisol (a cyclodextrin derivate used to solubilize carfilzomib)
* No macular degeneration or retinopathy (diabetic or otherwise) as examined during screening, or known porphyria or psoriasis (with the exception of early dry age-related macular degeneration or minor microhemorrhages in the retinal periphery)
* Well-controlled psoriasis allowed under care of a specialist who agrees to monitor the patient for exacerbations
* No other condition that would require therapy with hydroxychloroquine, including but not limited to, any of the following:
* Systemic lupus erythematosus
* Rheumatoid arthritis
* Porphyria cutanea tarda
* Malaria treatment or prophylaxis
* No concurrent or prior malignancy except for the following:
* Basal cell or squamous cell carcinoma of the skin
* Treated carcinoma in situ
* Localized prostate adenocarcinoma (stage T1a or T1b) with a stable prostate-specific antigen (PSA) for a period fo at least 4 months allowed
* Patients with a prior malignancy treated with chemotherapy, biologic agents, and/or radiation are eligible for this study if they have completed therapy ≥ 2 years previously with no evidence of recurrent disease
* Patients with a prior malignancy treated with surgery alone are eligible for this study if they have completed therapy ≥ 2 years previously with no evidence of recurrent disease
* No uncontrolled intercurrent illness including, but not limited to, any of the following:
* Uncontrolled ongoing infection
* Known acute or chronic hepatitis B, active hepatitis A or C or human immunodeficiency virus (HIV)
* Symptomatic congestive heart failure, defined as New York Heart Association (NYHA) Class III or IV
* Unstable angina pectoris
* Myocardial infarction within 6 months of enrollment
* Cardiac arrhythmia
* Clinically significant pericardial disease
* Cardiac amyloidosis
* Severe lung disease
* Psychiatric illness or social situations that would prevent compliance with study requirements

Prior and concurrent therapy

* No prior dose reductions of carfilzomib administration in previous lines
* At least 14 days since prior antimyeloma agents, not including carfilzomib/dexamethasone
* Concurrent therapy with bisphosphonates allowed at the discretion of the treating physician
* Concurrent hematopoetic growth factors allowed, including filgrastim granulocyte colony-stimulating factor (G-CSF) or pegfilgrastim, epoetin alpha, and darbepoetin alpha
* Concurrent participation in non-treatment studies allowed, if it will not interfere with participation in this study
* No concurrent radiotherapy except local radiotherapy during the treatment phase of this study for palliation of pain or prevention of fracture
* No concurrent treatment with a different investigational regimen
* No concurrent treatment with other anticancer agents
* No concurrent participation in other investigational trials that involve novel therapies

Ethical/other

* Female patients of child-bearing potential (FCBP) must have negative serum pregnancy test within 21 days prior to registration and agree to use an effective method of contraception during and for 3 months following last dose of drug.
* Male patients must use an effective barrier method of contraception during study and for 3 months following the last dose if sexually active with a FCBP.
* Ability to understand and willingness to sign the informed consent document
* Signed informed consent and expected cooperation of the patients for the treatment and follow up must be obtained and documented according to International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use - Good Clinical Practice (ICH-GCP), and national/local regulations.

Exclusion Criteria:

* Not meeting inclusion criteria
* Female patients who are pregnant or lactating.
* Any reason why, in the opinion of the investigator, the patient should not participate (e.g. not able to comply with study procedures, including being unable to perform full ophthalmologic examination).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose of hydroxychloroquine when added to standard-dose regimen of carfilzomib/dexamethasone | 3 months

SECONDARY OUTCOMES:
estimate of toxicity rate of hydroxychloroquine when added at a maximum tolerated dose to standard-dose regimen of carfilzomib/dexamethasone | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Torstein Baade Rø, Study Director — NTNU Department of Clinical and Molecular Medicine (IKOM); Tobias S Slørdahl, MD PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (2):
- Norway (2):
  - Oslo University Hospital, Department of Hematology, Oslo Myeloma Center, Oslo
  - St. Olavs Hospital, Department of Hematology, Trondheim

IPD SHARING:
Plan to Share IPD: Yes
tba

REFERENCES:
- [Derived] Slordahl TS, Askeland FB, Hanssen MSS, Hov H, Sundt-Hansen SM, Lindahl S, Vethe NT, Hjorth-Hansen H, Fenstad MH, Waage A, Hjertner O, Schjesvold F, Sundan A. Combined Proteasome and Autophagy Inhibition in Relapsed/Refractory Multiple Myeloma-A Phase I Trial of Hydroxychloroquine, Carfilzomib, and Dexamethasone. EJHaem. 2025 Jan 23;6(1):e1091. doi: 10.1002/jha2.1091. eCollection 2025 Feb. PMID 39866949